CLINICAL TRIAL: NCT05984888
Title: Protecting the Brain From Toxic Side Effects of Chemotherapy: a Pilot Study of a MIND Diet Intervention in Women Undergoing Active Treatment for Breast Cancer
Brief Title: Pilot Study of a MIND Diet Intervention in Women Undergoing Active Treatment for Breast Cancer
Acronym: MIND-BC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Tonya Orchard, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-22367
Record Dates: First submitted 2023-05-17; First posted 2023-08-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIND-BC Intervention Group (Experimental): Individual, tailored, behaviorally based nutrition counseling provided by a Registered Dietitian Nutritionist (RDN) and dietetic interns.
  Interventions: Behavioral: MIND Diet Intervention Group
- General Health Curriculum (GHC) Control (Active Comparator): Sessions of non-diet related health topic education.
  Interventions: Behavioral: General Health Curriculum (GHC) Group

INTERVENTIONS:
Behavioral: MIND Diet Intervention Group — Participants will receive individually tailored nutrition counseling on adopting the MIND diet pattern from a registered dietitian nutritionist (RDN) for a total of 8 sessions spanning 12 weeks. After completing the counseling sessions participants will be followed up 6 months later to collect additional questionnaires and assessments.
  Arms: MIND-BC Intervention Group
Behavioral: General Health Curriculum (GHC) Group — Participants will meet with trained study staff for 8 sessions spanning 12 weeks covering content on non-diet related health topics. After these sessions, participants will be followed up 6 months later to collect additional questionnaires and assessments. Once 6-month follow-up has been completed, participants will be offered to receive the MIND diet intervention offered in the MIND Diet Intervention Group.
  Arms: General Health Curriculum (GHC) Control

SUMMARY:
Breast cancer (BC) is the most frequently diagnosed cancer in women. Systemic cancer treatments are an important contributor to dramatic improvements in the long-term survival of women with BC. However, cancer treatment can lead to cognitive impairment and declines in quality of life in women with BC. Many cancer survivors experience memory and brain function decline following chemotherapy which can last for years. A newer diet pattern, Mediterranean-DASH [Dietary Approaches to Stop Hypertension] Intervention for Neurodegenerative Delay (MIND), was shown to help with protecting brain functions. The MIND diet is high in anti-inflammatory nutrients (e.g., omega-3 polyunsaturated fatty acids (PUFAs), carotenoids, B-vitamins, and polyphenols) and limits the intake of brain-unhealthy foods (i.e., butter/margarine, cheese, red meat, fried foods, pastries, and sweets), which may help alleviate negative cognitive outcomes from cancer treatments. This randomized controlled trial aims to investigate the effect of the MIND diet on cognitive functions in women with invasive BC starting systemic therapies.

ELIGIBILITY:
Inclusion Criteria:

* Stage II-IV hormone receptor+, breast cancer diagnosis
* Post-menopausal (defined as at least 1-year post menses, on ovarian suppression medication, or s/p oophorectomy)
* Within 4 weeks before or 12 weeks after starting initial systemic therapies (e.g. chemotherapy, targeted therapies such as CDK4/6 inhibitors, endocrine therapy)
* Ability to access and use internet resources, including video calls using Zoom platform
* English speaking

Exclusion Criteria:

* History of dementia, stroke, traumatic brain injury, brain metastasis or other conditions that could lead to cognitive impairment
* MIND diet score >8
* Unwilling/unable to eat >2 types of MIND food
* Receiving insulin therapy for diabetes
* Diagnosis of triple negative breast cancer
* Unable to give informed consent.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Remote Assessment of Cognition using the Hopkins Verbal Learning Test (HVLT) | One day
  Assess cognition remotely through a Zoom session by using the Hopkins Verbal Learning Test (HVLT), a brief cognitive test of episodic memory and verbal learning. The HVLT is broken down into three trials of free-recall from a 12-item list of words, followed by a period of time then a fourth recall trial. Finally, the test ends with a recognition task. For all trials, the maximum score is 12 with higher scores indicating better cognition.
Remote assessment of cognition using the WAIS-IV Digit Span | One day
  Assess cognition remotely through a Zoom session by using the Wechsler Adult Intelligence Scale (WAIS)-IV Digit Span, a cognitive test of attention and working memory. The WAIS-IV Digit Span is comprised of three individual tests: Digit Span Forward, Digit Span Backward, and Digit Span Sequence. A total potential score of 48 with higher scores indicating better cognition.
Remote assessment of cognition using the Oral Trail Making Test | One day
  Assess cognition remotely through a Zoom session by using the Oral Trail Making Test (TMT), a brief cognitive test of executive function and attention. The OTMT is divided into part A and part B. The part A asks participants to count from 1-25, while part B asks participants to alternate between letters and numbers. The less amount of time required to complete the task equates to better cognition.
Remote assessment of cognition using the COWA Test | One day
  Assess cognition remotely through a Zoom session by using the Controlled Oral Word Association (COWA) Test, a brief cognitive test of oral fluency and executive function. The COWAT has two components, the first asks the participants to say as many words as possible that begin with a given letter (F, A, or S) within the one-minute time frame. The second trial asks the same task but instead of letters, the participant is asked to produce as many animals as possible within the provided time frame. More words produced are indicative of better cognitive function.

SECONDARY OUTCOMES:
Assessment of presence of CRCI symptoms (Neuro-Qol) | One day
  Assess the presence of cancer-related cognitive impairment (CRCI) symptoms using the Neuro-QoL Cognitive Function Test, a self-report measurement of cognitive function. Higher scores indicate better cognitive functioning with a range from 8 - 40 for the raw score and a T-score range from 17.3 - 64.2.
Assessment of presence of CRCI symptoms (FACT-Cog) | One day
  Assess presence of cancer-related cognitive impairment (CRCI) symptoms using the Functional Assessment of Cancer Therapy - Cognition (FACT-Cog), a self-report measurement of cognitive function. Higher scores indicate better cognition with a range from 0 - 80.
Assessment of Diet Quality Measures | One day
  Assess diet quality measures from an electronic food frequency questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya S Orchard, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu